CLINICAL TRIAL: NCT02547220
Title: A Randomized Double-blind Placebo-controlled Study to Evaluate the Efficacy and Safety of Cinryze® (C1 Esterase Inhibitor [Human]) for the Treatment of Acute Antibody-mediated Rejection in Kidney Transplant Patients
Brief Title: A Multicenter Study to Evaluate the Efficacy and Safety of Cinryze® for the Treatment of Acute Antibody-mediated Rejection in Participants With Kidney Transplant
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Following a pre-scheduled interim analysis performed by the DMC, it was determined that the study met the pre-specified criteria for futility.
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SHP616-302; 2015-000726-11 (EudraCT Number)
Record Dates: First submitted 2015-09-02; First posted 2015-09-11 (Estimated); Results first posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-05

CONDITIONS: Acute Antibody-Mediated Rejection (AMR)
MeSH Terms: interventions — SERPING1 protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cinryze® (Experimental): Participants will receive 5000 Units of CINRYZE (50 millilitre [mL] of CINRYZE/ 50 mL of normal saline) on Day 1 and 2500 Units of CINRYZE (25 mL of CINRYZE/ 75 mL of normal saline) on Day 3, 5, 7, 9, 11, and 13 respectively.
  Interventions: Biological: Cinryze®
- Placebo (Placebo Comparator): Participants will receive 7 doses of matched placebo over 13 days of treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Cinryze® — Participants will receive 5000 Units of CINRYZE (50 millilitre [mL] of CINRYZE/ 50 mL of normal saline) on Day 1 and 2500 Units of CINRYZE (25 mL of CINRYZE/ 75 mL of normal saline) on Day 3, 5, 7, 9, 11, and 13 respectively.
  Arms: Cinryze®
Drug: Placebo — Participants will receive 7 doses of matched placebo over 13 days of treatment.
  Arms: Placebo

SUMMARY:
The main purpose of the study is to evaluate the efficacy of CINRYZE administered with plasmapheresis, plasma exchange, or immune adsorption treatments and sucrose-free immunoglobulin (IVIg) for the treatment of acute antibody-mediated rejection (AMR) of renal allograft in kidney transplant recipients as measured by the proportion of participants with new or worsening transplant glomerulopathy (TG) at 6 months after treatment initiation.

ELIGIBILITY:
Inclusion Criteria:

1. Be greater than or equal to (>=) 18 and less than or equal to (<=) 70 years of age.
2. Weigh >= 45 kg with a body mass index (BMI) less than (<) 35 kilogram (kg)/meter (m)^2 at screening.
3. Have human leukocyte antigen (HLA) donor-specific antibody (DSA) identified at the time of diagnosis of AMR. If it is anticipated that the local DSA results will not be available within the screening period, previously obtained local DSA results can be used to assess eligibility, if obtained after kidney transplant and within 30 days prior to the qualifying AMR episode. In any instance, a local DSA test should still be performed at the time of AMR diagnosis.
4. Have a first qualifying episode of AMR in the participant's current renal allograft between 72 hours (h) and 12 months after transplant defined by a renal allograft biopsy demonstrating neutrophil and/or monocyte infiltration in the peritubular capillaries (PTC) and/or glomeruli with or without evidence of 4th complement protein degradation product (C4d) deposition by immunohistopathology according to 2013 Banff criteria.
5. Have achieved adequate renal function defined as: Pre-AMR baseline estimated glomerular filtration rate calculated by the Modification of Diet in Renal Disease (eGFRMDRD) >=20 millilitre (mL)/minute (min) /1.73m^2 for a qualifying AMR episode occurring <=21 days after transplant or pre-AMR baseline eGFRMDRD >=30 mL/min/1.7m^2 for a qualifying AMR episode occurring greater than (>) 21 days after transplant. The pre-AMR baseline is the highest eGFRMDRD value obtained following the kidney transplant and within 30 days prior to the qualifying AMR episode. If more than 1 eGFRMDRD value is available, a mean of the 2 highest values (at least 1 day apart and both prior to the AMR episode) will be used as the pre-AMR baseline value. If no eGFRMDRD was obtained within 30 days prior to biopsy, it can be evaluated within a 60 day period.
6. Receive first dose of investigational product after 7 days after the kidney transplant procedure and within 7 days after the qualifying renal allograft biopsy procedure that was positive for AMR.
7. Be informed of the nature of the study and provide written informed consent before any study-specific procedures are performed.
8. If female and of child-bearing potential, must have a negative urine pregnancy test confirmed by a negative serum beta human chorionic gonadotropin (beta-HCG) pregnancy test at the Screening Visit and must have a negative urine pregnancy test at the Day 1 visit.
9. Agree to comply with any applicable contraceptive requirements of the protocol.

Exclusion Criteria:

1. Have received pediatric en bloc kidney transplant.
2. Have primary Focal Segmental Glomerulosclerosis, rapidly progressive glomerulonephritis, membrano-proliferative glomerulonephritis type 1 (including C3 glomerulopathy), "dense deposit disease", or thrombotic microangiopathy as the cause of native kidney failure.
3. Have prior or concurrent non-renal solid organ transplant or hematopoietic stem cell transplant (HSCT) or have more than 2 completed kidney transplant procedures (note: 1 double kidney transplant procedure is considered to be 1 procedure).
4. Have a known neoplastic lesion in the transplanted allograft
5. Have, any ongoing infection that causes hemodynamic compromise or as determined by the investigator, any surgical or medical condition that could interfere with the administration of investigational product, interpretation of study results, or could compromise participant safety, including (as determined by the transplanting surgeon and documented in the operative report) any major technical complications of the renal artery, renal vein, or ureteral anastomosis
6. Have ongoing treatment for hepatitis C virus (HCV) infection.
7. Have had a recent myocardial infarction (MI) within the past 6 months and/or at the time of screening are treated with anticoagulants and/or antiplatelet agents (excluding aspirin) for a previous myocardial infarction.
8. Have a history of: abnormal bleeding, clotting events or disorders (excluding a history of clotted hemodialysis access or superficial thrombophlebitis in the absence of medically confirmed coagulopathy), any coagulopathy (documented or clinically suspected) For example, participants should be excluded if they have a history of renal allograft arterial or venous thrombosis, deep vein thrombosis, pulmonary embolism, ischemic cerebrovascular accident (stroke) or transient ischemic attack (TIA), any large vessel thrombosis.
9. Have a history of allergic reaction to CINRYZE or other blood products.
10. Have had any change in androgen therapy (example, danazol, oxandrolone, stanozolol, testosterone), tranexamic acid, epsilon-aminocaproic acid, or other fibrinolytics within 3 months before the first dose of investigational product.
11. Have participated in the active dosing phase of any other investigational drug study within 30 days prior to dosing with investigational product.
12. Have any of the following local laboratory values reported prior to dosing with investigational product: Within 24 h prior to participant dosing, white blood cell (WBC) count <0.5×109/litre (L) or >20×109/L (the value of >20×109/L should be excluded if obtained during steroid treatment), Within 24 h prior to participant dosing platelet count <25×109/L or >600×109/L
13. Be pregnant or breastfeeding.
14. Have received any of the following agents within 1 month prior to the first dose of investigational product: Sucrose-containing intravenous immunoglobulin (IVIg), Any C1 inhibitor (C1 INH) (plasma-derived [example, CINRYZE®, Berinert®, Cetor®] or recombinant [example, Rhucin®]), Eculizumab (Soliris®), Ecallantide (Kalbitor®).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-05-20 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (47):
- United States (29):
  - Kidney Transplant Research Office at UCLA, Los Angeles, California
  - Keck School of Medicine at USC, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - University Of Colorado School Of Medicine, Aurora, Colorado
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Jackson Memorial Hospital, Miami, Florida
  - Florida Hospital Transplant Institute, Orlando, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Brigham and Womens Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Mount Sinai Hospital, New York, New York
  - Columbia University Medical Center, New York, New York
  - New York Presbyterian Hospital - Weill-Cornell, New York, New York
  - NYU Longone Medical Center, White Plains, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - INTEGRIS Nazih Zuhdi Transplant Institute, Oklahoma City, Oklahoma
  - University of Pittsburgh Medical Center, Monroeville, Pennsylvania
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor All Saints Medical Center, Fort Worth, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah
- Canada (2):
  - Providence Health Care Research Institute, Vancouver, British Columbia
  - Royal Victoria Hospital, Montreal, Quebec
- France (7):
  - Hotel Dieu, Nantes, Loire-Atlantique
  - Hopital Henri Mondor, Créteil, Val-De-Marne
  - CHU Michallon, Grenoble
  - Centre Hospitalier Universitaire de Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Saint Louis, Paris
  - Groupe Hospitalier Necker Enfants Malades, Paris
  - Hôpital de Rangueil, Toulouse
- Germany (3):
  - Universität Heidelberg, Heidelberg, Baden-Wurttemberg
  - Universitätsklinikum Frankfurt, Steinbach, Hesse
  - Universitätsklinikum Hamburg Eppendorf, Hamburg
- Netherlands (2):
  - Universitair Medisch Centrum Groningen, Groningen
  - Erasmus MC, Rotterdam
- Spain (4):
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Shire provides access to the de-identified individual participant data for eligible studies to aid qualified researchers in addressing legitimate scientific objectives. These IPDs will be provided following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.shiretrials.com website. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://www.shiretrials.com/en/our-commitment-to-transparency/data-sharing-with-researchers

REFERENCES:
- [Derived] Karpman D, Bekassy Z, Grunenwald A, Roumenina LT. A role for complement blockade in kidney transplantation. Cell Mol Immunol. 2022 Jul;19(7):755-757. doi: 10.1038/s41423-022-00854-5. Epub 2022 Mar 24. No abstract available. PMID 35332298

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 49 sites between 20 May 2016 (first participant first visit) and 31 May 2019 (last participant last visit).
Pre-assignment Details: A total of 39 participants were randomized and received treatment.
Groups:
- Placebo: Participants received a total of seven doses with an initial 100 mL intravenous (IV) infusion containing 5000 units of placebo (100 mL 0.9 percent [%] sodium chloride) on day 1 followed by 2500 units of placebo (100 mL 0.9% sodium chloride) on Days 3, 5, 7, 9, 11, and 13.
- CINRYZE: Participants received a total of seven doses with an initial 100 mL intravenous (IV) infusion containing 5000 units of CINRYZE on Day 1 followed by 2500 units of CINRYZE in 100 mL of IV infusion on Day 3, 5, 7, 9, 11, and 13.
Period: Overall Study
Arm/Group | Placebo | CINRYZE
Started | 19 | 20
Completed | 0 | 0
Not Completed | 19 | 20
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Study terminated by sponsor | 18 | 20

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) consisted of all participants who had taken at least 1 dose of investigational product.
Groups:
- Placebo: Participants received a total of seven doses with an initial 100 mL intravenous (IV) infusion containing 5000 units of placebo (100 mL 0.9% sodium chloride) on day 1 followed by 2500 units of placebo (100 mL 0.9% sodium chloride) on Days 3, 5, 7, 9, 11, and 13.
- Total: Total of all reporting groups
Arm/Group | Placebo | CINRYZE | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.9 (12.49) | 49.2 (13.45) | 50.5 (12.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 14
  Male | 10 | 15 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 9
  Not Hispanic or Latino | 13 | 10 | 23
  Unknown or Not Reported | 3 | 4 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 12 | 13 | 25
  American Indian or Alaska Native | 0 | 0 | 0
  Asian/Non-Japanese | 5 | 1 | 6
  Asian/Japanese | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 2 | 2 | 4
  Latino | 0 | 1 | 1
  Unknown | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With New or Worsening Transplant Glomerulopathy (TG) at Month 6 Post-Treatment
Description: New or worsening TG at month 6 by the standard score was defined as an increase in one or more between qualifying biopsy and 6-month biopsy. New or worsening TG was measured by Banff 2013 criteria (standard score) using allograft glomerulopathy (Cg0-Cg3): Cg0- No GBM double contours by light microscopy (LM) or electron microscopy (EM); Cg1- no GBM double contours by LM but GBM double contours in at least 3 glomerular capillaries by EM; Cg2- Double contours affecting 26 to 50% of peripheral capillary loops in the most affected of nonsclerotic glomeruli; Cg3- Double contours affecting more than 50% of peripheral capillary loops in the most affected of nonsclerotic glomeruli with a score range of 0 (no allograft glomerulopathy) and 3 (severe glomerulopathy). Percentage of participants with new or worsening TG at Month 6 post-treatment was reported.
Time Frame: Month 6
Population: FAS consisted of all participants who had taken at least 1 dose of investigational product.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | CINRYZE
Number analyzed (Participants) | 19 | 20
Percentage of participants | 47.4 | 50.0
Statistical Analysis 1: Comparison: Placebo vs CINRYZE; Test type: Superiority; p = 0.6857, Fisher Exact; Difference in percentage = 2.6, 95% CI 2-sided [-29.4 to 34.5] — Difference in percentage was calculated by the difference in percentage of new or worsening TG at 6 months between CINRYZE and placebo

2. Secondary Outcome: Number of Participants With All-Cause Graft Failure at Month 48
Description: Graft failure was determined as the presence of one or more of the following criteria: institution of permanent dialysis (defined as dialysis treatment more than [>] 30 days), current transplant nephrectomy, and/or a clinical determination of cessation of kidney graft function and estimated glomerular filtration rate (eGFR) less than or equal to (<=) 15 milliliter (mL)/minute (min)/1.73 meter (m)^2.
Time Frame: Month 48
Population: This study was prematurely terminated at Month 36 due to futility issue. This outcome measure was planned to analyze at Month 48. Hence, data for this outcome measure was not collected as planned, analyzed and reported.
Arm/Group | Placebo | CINRYZE
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change From Baseline in Renal Function up to Month 48
Description: Renal function was measured as glomerular filtration rate calculated by the modification of diet in renal disease (eGFRMDRD).
Time Frame: Baseline, up to Month 48
Population: as for outcome 2
Arm/Group | Placebo | CINRYZE
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change From Baseline With Pre-Antibody-Mediated Rejection (AMR) in Renal Function up to Month 48
Description: Renal function was measured as glomerular filtration rate calculated by the modification of diet in renal disease (eGFRMDRD). Pre-AMR baseline was the highest eGFRMDRD value obtained following the kidney transplant and within 30 days prior to the qualifying AMR episode.
Time Frame: Pre-AMR Baseline, up to Month 48
Population: as for outcome 2
Arm/Group | Placebo | CINRYZE
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Participants With Proteinuria Levels at Month 48
Description: Proteinuria included spot urine protein, urine creatinine, and urine protein/urine creatinine ratio.
Time Frame: Month 48
Population: as for outcome 2
Arm/Group | Placebo | CINRYZE
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change From Pre-Antibody-Mediated Rejection (AMR) Baseline in Histopathology Per Banff Criteria at Month 6
Description: Histopathological diagnosis of acute rejection was measured by Banff 2013 criteria: Glomerulitis score (g0-g3), allograft glomerulopathy (Cg0-cg3), Tubulitis score (T0-T3), Intimal arteritis score (V0-V3), peritubular capillaritis (PTC) (ptc0-ptc3) and Interstitial Inflammation score (i0-i3). The histopathology was a composite of the sub-scores. Each of the sub-scores or histopathology score ranges from 0 ( no histopathology) to 3 (more severe histopathology).
Time Frame: Pre-AMR Baseline, Month 6
Population: This study was prematurely terminated at Month 36 due to futility issues. The data of this secondary outcome measure was not collected as planned and the secondary analysis was not performed, due to early study termination.
Arm/Group | Placebo | CINRYZE
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Number of Participants With All-Cause Graft Failure at Month 6
Description: Graft failure was determined by the presence of one or more of the following criteria: institution of permanent dialysis (defined as dialysis treatment more than [>] 30 days), current transplant nephrectomy, and/or a clinical determination of cessation of kidney graft function and estimated glomerular filtration rate (eGFR) less than or equal to (<=) 15 milliliter (mL)/minute (min)/1.73 meter (m)^2.
Time Frame: Month 6
Population: as for outcome 6
Arm/Group | Placebo | CINRYZE
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Number of Participants With Graft Failure Due to Antibody-Mediated Rejection (AMR) Episodes at Month 48
Description: as for outcome 7
Time Frame: Month 48
Population: as for outcome 2
Arm/Group | Placebo | CINRYZE
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Time to All-Cause Graft Failure up to Month 48
Description: Graft failure was determined by the presence of one or more of the following criteria: institution of permanent dialysis (defined as dialysis treatment more than [>] 30 days), current transplant nephrectomy, and/or a clinical determination of cessation of kidney graft function and estimated glomerular filtration rate (eGFR) less than or equal to (<=) 15 milliliter (mL)/minute (min)/1.73 meter (m)^2. Time to all-cause graft failure in months was calculated as (Date of graft failure - Date of first dose + 1)/30.25.
Time Frame: Up to Month 48
Population: as for outcome 2
Arm/Group | Placebo | CINRYZE
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Time to Graft Failure Due to Antibody-Mediated Rejection (AMR) Episodes up to Month 48
Description: Graft failure was determined by the presence of one or more of the following criteria: institution of permanent dialysis (defined as dialysis treatment > 30 days), current transplant nephrectomy, and/or a clinical determination of cessation of kidney graft function and eGFR <=15 mL/ min/1.73m^2. Time to graft failure due to AMR episodes in months was calculated as (Date of graft failure due to AMR - Date of first dose + 1)/30.25.
Time Frame: Up to Month 48
Population: as for outcome 2
Arm/Group | Placebo | CINRYZE
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Number of Participants With Resolution of the Qualifying Antibody-Mediated Rejection (AMR) Episodes at Month 48
Description: Number of participants with resolution of the qualifying AMR episodes at Month 48.
Time Frame: Month 48
Population: as for outcome 2
Arm/Group | Placebo | CINRYZE
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Time to Resolution of Qualifying Antibody-Mediated Rejection (AMR) Episodes up to Month 48
Description: Time to resolution of qualifying AMR episodes was calculated as (Date of qualifying AMR resolution - Date of first dose + 1)/30.25. Participants who didn't had resolution of qualifying AMR episodes and still on-study were censored at the date of last visit; Participants who had completed the study without resolution of qualifying AMR were censored at the date of study completion; participants who discontinued from the study without resolution of qualifying AMR were censored at the date of early discontinuation.
Time Frame: Up to Month 48
Population: as for outcome 2
Arm/Group | Placebo | CINRYZE
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Number of Participants Who Were Alive at Month 36
Description: Number of participants who were alive at Month 36 (study terminated instead of Month 48) were reported.
Time Frame: Month 36
Population: Safety analysis set consisted of all participants who had taken at least 1 dose of investigational product. This study was prematurely terminated at Month 36 due to futility issue. This outcome measure was planned to analyze at Month 48.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | CINRYZE
Number analyzed (Participants) | 19 | 20
Participants | 19 | 20

14. Secondary Outcome: Time to All-Cause Mortality up to Month 48
Description: Time to all-cause mortality was calculated as (Date of discontinuation due to death - Date of first dose + 1)/30.25. Participants who are alive and still on-study were censored at the date of last visit; Participants who had completed the study were censored at the date of study completion; Participants who discontinued from the study but not due to death were censored at the date of early discontinuation.
Time Frame: Up to Month 48
Population: as for outcome 2
Arm/Group | Placebo | CINRYZE
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward, undesired, unplanned clinical event in the form of signs, symptoms, disease, or laboratory or physiological observations occurred in a participant participating in a clinical study with the sponsor's product, regardless of causal relationship. TEAEs were defined as events that started or worsened on or after the date of the first dose of investigational product, but no later than 30 days following the last dose of investigational product, within a treatment period.
Time Frame: From start of study drug administration up to study termination (Month 36)
Population: Safety analysis set consisted of all participants who had taken at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | CINRYZE
Number analyzed (Participants) | 19 | 20
Participants | 16 | 16

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to study termination (Month 36)
Arm/Group | Placebo | CINRYZE
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 6/19 | 3/20
Other Adverse Events (participants affected / at risk) | 15/19 | 16/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=19) | CINRYZE (N=20)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Catheter site thrombosis (General disorders) | 0 (0) | 1 (1)
Anaphylactic shock (Immune system disorders) | 1 (1) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=19) | CINRYZE (N=20)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (3) | 1 (2)
Lymphocele (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tooth disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 2 (2) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Nodule (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 2 (2) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
BK virus infection (Infections and infestations) | 1 (1) | 0 (0)
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Arteriovenous fistula site haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Citrate toxicity (Injury, poisoning and procedural complications) | 0 (0) | 1 (5)
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood bicarbonate decreased (Investigations) | 0 (0) | 1 (1)
Blood bicarbonate increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0)
Blood magnesium decreased (Investigations) | 1 (1) | 0 (0)
Blood phosphorus decreased (Investigations) | 0 (0) | 1 (1)
Blood potassium increased (Investigations) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 1 (1) | 0 (0)
Blood uric acid increased (Investigations) | 1 (1) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 2 (2) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Folate deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (3) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was prematurely terminated at Month 36 due to futility issue.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2017-11-22): https://cdn.clinicaltrials.gov/large-docs/20/NCT02547220/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-27): https://cdn.clinicaltrials.gov/large-docs/20/NCT02547220/SAP_001.pdf